CLINICAL TRIAL: NCT07129590
Title: TRauma-Informed Care in Smoking cEssation for Pregnancy (RISE Pregnancy)
Brief Title: Trauma-Informed Care for Smoking Cessation for Pregnancy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Tobacco Related Disease Research Program (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 25634; NCI-2025-05151 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2025-08-11; First posted 2025-08-19 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Smoking Cessation; Tobacco Smoking; Tobacco Use Cessation; Smoking Reduction; Smoking, Cigarette; Trauma, Psychological; Trauma and Stressor Related Disorders
Keywords: Pregnancy
MeSH Terms: conditions — Smoking Cessation; Tobacco Smoking; Tobacco Use Cessation; Smoking Reduction; Cigarette Smoking; Psychological Trauma; Trauma and Stressor Related Disorders | interventions — Interviews as Topic; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aim 1: Development, Pilot Group (Experimental): Both clinician- and patient-participants will participate in a 60-minute in-depth, semi-structured interview conducted either in-person or via secure University of California, San Francisco (UCSF) video-telephone software.
  Interventions: Other: Expired carbon monoxide (CO); Other: Interviews; Other: Questionnaires

INTERVENTIONS:
Other: Expired carbon monoxide (CO) — Expired CO will be measured using a non-investigational device
  Other Names: Exhaled CO
Other: Interviews — Participants will be interviewed via video conference or in person
  Other Names: Participant Interviews
Other: Questionnaires — Participants will receive questionnaires to complete through the course of the study
  Other Names: Surveys

SUMMARY:
Trauma-informed approaches have been shown to support recovery from other substance use disorders and involve four key elements: (1) Realizing the prevalence of trauma and pathways to recovery, (2) Recognizing symptoms of trauma, (3) Responding by embedding knowledge of trauma into practices and policies and (4) Resisting re-traumatization (the 4Rs). In close partnership with Breathe California and a public safety-net clinic in San Francisco that serves primarily racial and ethnic minoritized (REM) pregnant women, the 4Rs along with the Ask, Advise, Assess, Assist and Arrange (the 5As) evidence-based intervention for tobacco cessation that is delivered by health care professionals and is a US Public Health Services clinical practice guideline for treating tobacco will be used to create and implement a smoking cessation intervention for pregnant women with experiences of trauma.

DETAILED DESCRIPTION:
This study is currently enrolling for Aim 1 only.

Study Objectives:

Aim 1: Assess barriers to successful maternal tobacco cessation for women with trauma and identify targets for intervention through interviewing pregnant women with trauma and clinicians in the safety-net using the Behavior Change Wheel (BCW), a validated implementation science behavior change framework.

Aim 2: Evaluate and adapt an evidence-based tobacco cessation intervention using the for pregnant women by incorporating trauma-informed approaches (the 4Rs) with the established 5As. Input will lead to the effective adaptation and creation of the final TRauma-Informed Care in Smoking cEssation for Pregnancy (RISE) Pregnancy intervention to be tested in Aim 3.

Aim 3: Determine the feasibility and acceptability of the RISE Pregnancy intervention and protocol.

OUTLINE:

This study is currently enrolling for Aim 1 only.

Aim 1: Pregnant women in the safety-net who smoke and have histories of trauma, and clinicians will be interviewed using the BCW to assess barriers to smoking cessation and inform design of a smoking cessation intervention which will be used to inform the design of a smoking cessation intervention (RISE Pregnancy) for evaluation in Aim 2.

ELIGIBILITY:
Inclusion Criteria:

Clinician Eligibility Criteria (Aims 1 - 3):

In Aims 1-3, will be recruiting clinicians working in the Obstetrics, Midwifery, and Gynecology Clinic (5M) safety-net clinic and the UCSF Community and Clinical Research Center (ZSFG).

1. Nurse practitioner, physician assistant, nurse-midwife, or medical doctor caring for pregnant patient-participants.
2. Age ≥ 18 years old.

Patient-participant Eligibility Criteria (Aim 1):

In Aim 1, will be recruiting pregnant women receiving care at the 5M safety-net clinic who are actively smoking and have histories of trauma (ages 18+)

1. Currently smoking
2. Age ≥18 years old.
3. Currently Pregnant.
4. Identifies as a cisgender woman, or female at birth.
5. Reports having experienced trauma aligned with Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) definition for traumatic exposure.
6. Proficient in English or Spanish languages.

Patient-Participant Eligibility Criteria (Aim 2):

Patient-participants from the 5M advisory boards will be recruited to give feedback on our intervention using Evidence-Based Quality Improvement (EBQI) meetings.

Inclusion criteria:

1. Participant in a 5M Clinic Patient Advisory Board.
2. Age ≥18 years old.
3. Proficient in English or Spanish languages.

Patient-Participant Eligibility Criteria (Aim 3): In Aim 3, will be recruiting pregnant women receiving care at the 5M safety-net clinic who are actively smoking and have histories of trauma (ages 18+).

Inclusion criteria:

1. Currently smoking (ever smoked 100 cigarettes in their lifetime, smoked in the past 7 days and at least 1 cigarette per day, verified by CO≥6ppm)
2. ≥18 years old
3. Currently Pregnant
4. Identifies as a cisgender women, or female at birth
5. Meets DSM-5 Criterion A for trauma exposure on the Brief Trauma Questionnaire (BTQ)
6. English or Spanish Proficient

Exclusion Criteria:

Clinician- and Patient-participant Exclusion criteria (Aims 1 - 3):

1. Any condition, including active mental health crises or cognitive impairment, that would interfere with the ability to provide informed consent or safely complete the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-11-19 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of themes (Aim 1) | Up to 6 months
  Themes related to how to improve smoking cessation for pregnant people will be identified through in-depth interviews.

CONTACTS AND LOCATIONS:
Overall Officials: Anita Hargrave-Bouagnon, MD, MAS, Principal Investigator — University of California, San Francisco
Locations (1):
- Zuckerberg San Francisco General Hospital, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No